CLINICAL TRIAL: NCT00180193
Title: F-18-OMFD-PET for Radiotherapy Treatment Planning and Evaluation of Early Therapy Response
Status: Terminated | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: Advanced Biochemical Compounds GmbH (Industry)
Responsible Party: Prof. Dr. med. Jörg Kotzerke, Klinik und Poliklinik für Nuklearmedizin
Other Study IDs: ABX-OMFD-FU
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Brain Tumor
Keywords: Radiotherapy; F-18-OMFD
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to monitor the amino acid uptake of brain tumors, before and during radiotherapy, with positron emission tomography.

ELIGIBILITY:
Inclusion Criteria:

* Brain tumor
* Radiation therapy indicated
* Written consent

Exclusion Criteria:

* Pregnancy
* Mental impairment
* Drug/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OMFD-PET of all patients after subtotal resection or biopsy of malignant glioma was evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Kotzerke, MD, Principal Investigator — Department of Nuclear Medicine
Locations (1):
- Department of Nuclear Medicine, Dresden, Germany